CLINICAL TRIAL: NCT01301118
Title: Split Thickness Skin Graft Take and Microbiology Evaluation in Burned Patients
Brief Title: Graft Take and Microbiology in Burns
Status: Suspended | Type: Observational
Why Stopped: Technical problems with protocol.
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, ALFREDO GRAGNANI FILHO, Associated Professor, Federal University of São Paulo
Other Study IDs: Graft take in burns
Record Dates: First submitted 2011-02-22; First posted 2011-02-23 (Estimated); Last update posted 2012-01-10 (Estimated); Status verified 2012-01

CONDITIONS: Transplantation Infection; Wound of Skin; Burns; Graft Loss; Infection
Keywords: Transplantation Infection; Wound of skin; Burns; Graft Loss; Infection
MeSH Terms: conditions — Burns; Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
SPLIT-THICKNESS SKIN GRAFT TAKE AND MICROBIOLOGICAL EVALUATION IN BURNED PATIENTS

INTRODUCTION: Infection is cause of increased morbidity and mortality in burn patients, and its control is a major challenge also for skin graft integration. Wound and soft tissue infection rates are higher than microbiological diagnosis rates.

PURPOSE: To evaluate partial skin graft integration in relation to microbiological analysis of wounds in burn patients.

METHODS: This project will be a transversal, prospective, analytical, controlled study in humans, conducted in a single center, at Burn Care Unit of Department of Plastic Surgery at Federal University of São Paulo from October, 2010 to October, 2011. Data will be collected to characterize demographic and clinical aspects. Data analysis will be performed using Student's t-test and Friedman analysis of variance.

DETAILED DESCRIPTION:
SPLIT-THICKNESS SKIN GRAFT TAKE AND MICROBIOLOGICAL EVALUATION IN BURNED PATIENTS

INTRODUCTION: Early excision and partial skin graft is state-of-the-art in burns treatment. Otherwise, infection is cause of increased morbidity and mortality in burn patients, and its control is a major challenge also for skin graft integration. Wound and soft tissue infection rates are higher than microbiological diagnosis rates. This difference is related to moderate sensibility of cultures in general. Precise bacterial diagnostic and its susceptibility to specific antibiotics are prerequisite for adequate treatment of burn patients and skin graft integration.

PURPOSE: To evaluate partial skin graft integration in relation to microbiological analysis of wounds in burn patients.

METHODS: This project was approved at Ethics Committee at Federal University of São Paulo (1272/10). It will be a transversal, prospective, analytical, controlled study in humans, conducted in a single center, at Burn Care Unit of Department of Plastic Surgery at Federal University of São Paulo from October, 2010 to October, 2011. Thirty patients will be included in this study after reading and signing a consent form. Data will be collected using an evaluation sheet to characterize demographic and clinical aspects, including partial skin graft integration, use of topical and systemic antibiotics and infection rates in all sites (blood, urine, skin, tracheal aspirate and bronchial lavage). Data analysis will be performed using Student's t-test and Friedman analysis of variance.

ELIGIBILITY:
Inclusion Criteria:

* Both gender
* More than 18 years of age
* Burned patient
* Inpatient of Burn Center of Federal University of São Paulo
* Upper 5% of TBSA
* Debridement and skin graft indication and procedure realization

Exclusion Criteria:

* Not interest in participating in research
* Not have debridement or graft indication
* Under 5% of TBSA
* Skin disease
* Clinical disease that contraindication procedure
* Clinical disease that directly interferes with infectious process and wound healing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ACUTE BURNED PATIENTS
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2010-10

CONTACTS AND LOCATIONS:
Overall Officials: ALFREDO GRAGNANI, MD PhD, Principal Investigator — UFSaoPaulo; LYDIA M FERREIRA, MD Full Prof, Study Chair — UFSaoPaulo